CLINICAL TRIAL: NCT04931329
Title: Impact of an Onco-haematology Vigilance Card in the Optimisation of the Town-hospital Relationship.
Brief Title: Onco-haematology Vigilance Card
Acronym: THERANOVA-LIM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI21_0010
Record Dates: First submitted 2021-05-10; First posted 2021-06-18 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-07

CONDITIONS: Medical Oncology; Hematology; Molecular Targeted Therapies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to show the interest of setting up a drug vigilance card in Oncology in order to reinforce patient safety, develop compliance and avoid drug interactions when the patient consults town professionals or other specialists.

DETAILED DESCRIPTION:
Recent developments in oral chemotherapy and targeted therapies have radically changed cancer patient management; ambulatory care is now common. Oral therapies afford many advantages, improving patient quality of life and autonomy by reducing hospital stays and involving patients in their own care. Optimising the care of cancer patients at home requires the coordinated intervention of hospital and town healthcare professionals and involvement of the patient to detect, prevent, and manage adverse events, avoid drug interactions, and educate patients. Preliminary work in haematology has highlighted (n = 31 patients) the interest of a "drug vigilance card" in three indications (Chronic Lymphocytic Leukaemia, Chronic Myeloid Leukaemia and Multiple Myeloma) with an increase in the town-hospital link.

This is an prospective cohort study. Following the announcement consultation, in addition to the personalised care plan, the information about the treatment will be contained in a drug monitoring card that will be given to the patient by the health professional (doctor or nurse). This drug monitoring card should be presented to the health professionals by the patient. During the entire period of treatment, the patient will have a card.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated at Limoges University Hospital in Medical Oncology department, receiving oral treatment (chemotherapy and/or targeted therapies)

Exclusion Criteria:

* All patients treated at Limoges University Hospital in Medical Oncology department, receiving hormone therapy or IV treatment only.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with onco-heamatologic disease treated with oral treatment (chemotherapy and/or targeted thérapies)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
measure patient satisfaction at 3 months | 3 months
  Patient satisfaction will be evaluated using IBM computer usability satisfaction questionnaires published by James R. Lewis (https://doi.org/10.1080/10447319509526110)

SECONDARY OUTCOMES:
Measurement of caregiver satisfaction | 3 months
  Caregiver satisfaction will be evaluated using IBM computer usability satisfaction questionnaires published by James R. Lewis (https://doi.org/10.1080/10447319509526110)
Measurement of compliance reported by the GIRERD questionnaire | 3 months
  patients will have to answer shorts questions on GIRERD* questionnaire to evaluate their Medication compliance to oral anticancer drugs.
  *X. Girerd, O. Hanon, K. Anagnostopoulos, C. Ciupek, J.J. Mourad, S. Consoli Assessment of antihypertensive compliance using a self-administered questionnaire: development and use in a hypertension clinic Presse Med, 30 (2001), pp. 1044-1048
Measuring the satisfaction of treating physicians and health professionals | 3 months
  Treating physicians ad health professionnals satisfaction will be evaluated using IBM computer usability satisfaction questionnaires published by James R. Lewis (https://doi.org/10.1080/10447319509526110)
Evaluate the use of the QR code by health professionals/carers | 3 months
  The use of the QR code with be evaluated by counting how many times it will be flashed during study period.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Limoges, Limoges, France

REFERENCES:
- [Derived] Boucheteil M, Leobon S, Baffert KA, Huet S, Darbas T, Le Brun-Ly V, Pestre J, Peyramaure C, Thuillier F, Venat L, Jost J, Touati M, Deluche E. [THERANOVA-LIM: Improving access to information on oral treatments for patients and pharmacists]. Bull Cancer. 2025 Dec 17:S0007-4551(25)00521-1. doi: 10.1016/j.bulcan.2025.10.005. Online ahead of print. French. PMID 41412846